CLINICAL TRIAL: NCT05764070
Title: Impact of Vagus Nerve Stimulation on Post-Aerobic Activity Recovery in Post Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Patients
Brief Title: Impact of Vagus Nerve Stimulation on Post-Aerobic Activity Recovery in Post SARS-CoV-2 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, physiotherapist PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SARS-CoV-2
Record Dates: First submitted 2023-03-09; First posted 2023-03-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Masking Description: Evaluation and treatment will be carried out by different physiotherapists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Invasive Vagus Stimulation (Experimental): Aerobic exercise + Non Invasive- Vagus Stimulation
  Interventions: Device: non-invasive auricular vagus stimulation
- Placebo Non Invasive Vagus Stimulation (Placebo Comparator): Aerobic exercise + Placebo Non Invasive Vagus Stimulation
  Interventions: Device: Placebo Non Invasive Vagus Stimulation

INTERVENTIONS:
Device: non-invasive auricular vagus stimulation — The only cutaneous nerve of the N. vagus, ramus auricularis, receives sensation from the posterior surface of the auricle, the posterior part of the external auditory canal and the adjacent part of the eardrum. Non-invasive transcutaneous devices stimulate the vagus nerve via the auricular route or from the carotid. This device non-invasively stimulates the auricular branch of the vagus nerve without any action. As a result, it was found that the pain threshold increased and the mechanical pain sensitivity decreased.
  Arms: Non Invasive Vagus Stimulation
Device: Placebo Non Invasive Vagus Stimulation — Placebo Non Invasive Vagus Stimulation
  Arms: Placebo Non Invasive Vagus Stimulation

SUMMARY:
Chronic fatigue, weakness, dyspnea, headaches, cognitive dysfunction, stress, sadness, anxiety, sleep disturbances, and orthostatic intolerance are among the symptoms of acute Covid-19 in patients, and these symptoms persist for more than 12 weeks after recovery. Extended Covid-19 syndrome, also known as Post-Covid-19 syndrome, is described as

DETAILED DESCRIPTION:
Therapeutic exercises are an evidence-based method for the maintenance of musculoskeletal, cardiovascular and neurological well-being and the prevention and treatment of chronic diseases. The effects of therapeutic exercises on the human body varied according to the frequency, intensity, duration and type of exercise.

Increasing physiological and psychological recovery after exercise can lead to results such as better performance and reducing the risk of injury. Therefore, various methods are used to facilitate post-exercise recovery.

The best-known and most widely used post-exercise recovery method is active cooling, also known as active rest or cool-down. Active cooling; It is defined as any activity that includes voluntary, low/moderate intensity exercise or movement performed within one hour of exercise. Passive rest, on the other hand, is defined as no or minimal voluntary/intentional exercise movement.

ELIGIBILITY:
Inclusion criteria:

* Covid
* be between 18-45 years old
* Having pulmonary involvement in the covid process

Exclusion criteria:

* Being a professional in any sport
* Having a cardiopulmonary, orthopedic, neurological and metabolic disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | a day
  In the measurement of pain intensity, it was planned to use a standard, 10 mm VAS with proven reliability. The severity of pain felt by the patient; It is a scale used to mark 0 = no pain and 10 = the most severe pain, thus determining the patient's pain intensity subjectively.
Autonomic nervous system device (Polar H10) | a day
  The Polar H10 device is a heart rate sensor that comes with a wearable chest strap and is the gold standard of high sensitivity and accuracy. It can be connected to multiple training devices via Bluetooth and ANT+. The device comes with a soft, adjustable sensor that touches the chest to capture the heart rate in real time.
  In the study, the autonomic nervous system will be evaluated with the Polar H10 device. By connecting the device to a smart phone via bluetooth, the data will be recorded and the software supported by the device will be used for the analysis of the data.
Lactate Analysis | one day
  It was measured with a portable lactate analyzer before and after exercise training, just before the recovery phase. It is an ideal lactate analyzer for using metabolic information to assess endurance, design optimal training programs, avoid overtraining plans and help identify target heart rate zones.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir University, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

REFERENCES:
- [Background] McNarry MA, Berg RMG, Shelley J, Hudson J, Saynor ZL, Duckers J, Lewis K, Davies GA, Mackintosh KA. Inspiratory muscle training enhances recovery post-COVID-19: a randomised controlled trial. Eur Respir J. 2022 Oct 6;60(4):2103101. doi: 10.1183/13993003.03101-2021. Print 2022 Oct. PMID 35236727